CLINICAL TRIAL: NCT01887132
Title: A Randomized Controlled Trial of Donepezil for REM Enhancement and Behavioral Change in Autism
Brief Title: A Trial of the Drug Donepezil for Sleep Enhancement and Behavioral Change in Children With Autism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130164; 13-M-0164
Record Dates: First submitted 2013-06-22; First posted 2013-06-26 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Autism Spectrum Disorders
Keywords: Sleep Architecture; Autism; Language Development
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Donepezil

ARMS (3):
- Open-Label Donepezil (Experimental)
  Interventions: Drug: Donepezil
- Donepezil - Blinded (Experimental)
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil
  Arms: Donepezil - Blinded; Open-Label Donepezil
Drug: Placebo
  Arms: Placebo

SUMMARY:
Background:

- Some children with autism spectrum disorders (ASD) do not have normal sleep cycles. Some of these children spend very little time in the rapid eye movement (REM) stage of sleep. Some studies suggest that less time in REM sleep can be associated with learning and behavior problems. Donepezil is a medication used to treat Alzheimer s disease. Donepezil can increase REM sleep in some adults with different disorders. A small study showed that Donepezil can also increase REM sleep in children with ASD. Researchers now want to see if Donepezil can improve communication skills and social interaction in children with ASD. They also want to see if any change in symptoms seems to come from changes in REM sleep.

Objectives:

- To see if a medication, Donepezil, can improve the way communication skills and social interaction develop in young children with autism spectrum disorders.

Eligibility:

- Children 22 to 44 months of age with ASD.

Design:

* Participants will be screened with a blood test, heart tests, and a sleep study. During the sleep study, children will sleep in a darkened room for 2 nights with electrodes on their body and a tube under their nose. Parents can sleep in the room with their child. A technician will monitor the room all night.
* Participants will take the study medication once a day.
* Treatment will be monitored at visits every 3 months. At each visit the participant will take blood tests, heart tests, or behavior tests. Participants will have 2 more sleep studies.
* Participation will end after 18 months.

DETAILED DESCRIPTION:
i. Objective

The objective of this study is to investigate the efficacy of donepezil to improve the developmental trajectory for core behavioral domains specific to autism, namely reciprocal social interaction and communication.

ii. Study population

90 children with an autism spectrum disorder between the ages of 24 to 50 months will be screened via polysomnogram to find 45 with a relative REM deficiency. This group will then be divided into two arms of drug versus placebo. Allowing for a 22 % drop out rate we expect 17 in each group to complete the study. Additionally, we will enroll 16 children with an ASD who do not meet criteria for relative REM deficiency in an open label arm to ascertain whether or not donepezil is beneficial to behavior in this group.

iii. Design

The proposal is for a 6 month treatment trial of 2.5 mg donepezil/placebo/day followed by 12 months of longitudinal follow-up. The primary study endpoint will be an examination of autism core symptoms and sleep architecture after 12 months.

iv. Outcome measures

The primary outcome measure will be:

1. An improvement in the Expressive Language and the Receptive Language subscales of the Mullen Scales of Early Learning (MSEL) at 12 months.

   Secondary outcome measures will be:
2. We will also measure the change in REM sleep parameters after 6, 12 and 18 months in relation to improvements in behavioral indices.

   Exploratory Outcome Measures will be:
3. An improvement in the Expressive Language and the Receptive Language subscales of the Mullen Scales at 18 months.
4. An improvement on the severity scale of the Autism Diagnostic Observation Schedule (ADOS) at 6, 12 and 18 months.
5. An improvement on the Vineland at 3, 6, 12 and 18 months
6. An exploratory analysis will investigate whether normalization of REM parameters also improves other measurements of sleep quality in children with autism.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis of an Autism Spectrum Disorder (DSM-IV diagnoses of autistic disorder or Pervasive Developmental Disorder, Not Otherwise Specified).
  2. Male or Female subjects between the ages of 24 and 50 months.
  3. Language scores (from the Mullen Scales of Early Learning) that are at least 1.5 SD lower than the mean.

  5. Each legal guardian must have a level of understanding sufficient to agree to all required tests and examinations. Each legal guardian must understand the nature of the study.

  6. Each subject must be stable for at least 6 weeks on any medication or therapy regimen prior to entry into study and must have no newly (within 6 weeks) recognized or intolerable adverse effects from that medicine or therapy. No subjects will be asked to discontinue any medication in order to qualify for enrollment but subjects taking contraindicated drugs will not qualify for enrollment.

  7. Demonstrated REM% two standard deviations or more below the normative values for age for the randomized controlled trial part.

  8. English language is primarily spoken at home.

EXCLUSION CRITERIA:

1. Serious, unstable illnesses including gastroenterologic, respiratory, cardiovascular endocrinologic, immunologic, or hematologic disease.
2. Renal or hepatic dysfunction that would interfere with excretion or metabolism of donepezil as evidenced by increase above upper limits of normal for BUN/creatinine, or two-fold elevation of serum transaminases (ALT/SGPT, AST/SGOT) or gamma glutamate (GGT).
3. Documented history of hypersensitivity or intolerance to donepezil or other piperidine derivative.
4. Subjects must not be taking any medication known to affect REM sleep (or sleep

   architecture in general) or that is contraindicated for co-administration with donepezil.
5. Presence or history of other unstable neurological disorders such as seizure disorders,

metabolic disorders, narcolepsy or movement disorders.

Ages: 24 Months to 50 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashura W Buckley, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD shared via NIMH repository protocol.

REFERENCES:
- [Background] Anderson DK, Lord C, Risi S, DiLavore PS, Shulman C, Thurm A, Welch K, Pickles A. Patterns of growth in verbal abilities among children with autism spectrum disorder. J Consult Clin Psychol. 2007 Aug;75(4):594-604. doi: 10.1037/0022-006X.75.4.594. PMID 17663613
- [Background] Anderson DK, Oti RS, Lord C, Welch K. Patterns of growth in adaptive social abilities among children with autism spectrum disorders. J Abnorm Child Psychol. 2009 Oct;37(7):1019-34. doi: 10.1007/s10802-009-9326-0. PMID 19521762
- [Background] Bliwise DL, Carroll JS, Lee KA, Nekich JC, Dement WC. Sleep and "sundowning" in nursing home patients with dementia. Psychiatry Res. 1993 Sep;48(3):277-92. doi: 10.1016/0165-1781(93)90078-u. PMID 8272449
- [Derived] Ure A, Cox GR, Haslam R, Williams K. Acetylcholinesterase inhibitors for autistic spectrum disorders. Cochrane Database Syst Rev. 2023 Jun 1;6(6):CD013851. doi: 10.1002/14651858.CD013851.pub2. PMID 37267443

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants signed consent. Only 4 started the study.
Groups:
- Open-Label Donepezil: Donepezil
Period: Overall Study
Arm/Group | Open-Label Donepezil
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Donepezil
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] — Mean age of the participants at screening.
  years | 3.2 [2.1 to 3.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Nonverbal Developmental Quotient (NVDQ)
Description: The Nonverbal Developmental Quotient (NVDQ) was calculated from the Mullen Scales of Early Learning scores by dividing the nonverbal mental age (average of the age equivalent value for the Visual Reception and Fine Motor scores) by the chronological age in months. The NVDQ is normalized to a mean score of 100, which indicates an average normal IQ. Less than 100 is a lower than average IQ. 2 standard deviations below average is considered "impaired" IQ (approximately lower than 70).
Time Frame: Baseline and 12 months
Measure: Number; unit: units on a scale
Arm/Group | Open-Label Donepezil
Number analyzed (Participants) | 4
units on a scale
  NVDQ for participant 1 at Baseline | 51.61
  NVDQ for participant 2 at Baseline | 48.89
  NVDQ for participant 3 at Baseline | 58.97
  NVDQ for participant 4 at Baseline | 54.88
  NVDQ for participant 1 at 12 mos | 52.38
  NVDQ for participant 2 at 12 mos | 44.74
  NVDQ for participant 3 at 12 mos | 54.00
  NVDQ for participant 4 at 12 mos | 45.45

2. Secondary Outcome: REM Percentage at Baseline, 6, 12 and 18 Months
Description: REM percentage is the percentage of sleep spent in REM
Time Frame: Baseline, 6, 12 and 18 months
Measure: Number; unit: percentage of sleep
Arm/Group | Open-Label Donepezil
Number analyzed (Participants) | 4
percentage of sleep
  REM percentage, participant 1, Baseline | 17.2
  REM percentage, participant 2, Baseline | 18.6
  REM percentage, participant 3, Baseline | 19.9
  REM percentage, participant 4, Baseline | 12.1
  REM percentage, participant 1, 6 mos | 27.5
  REM percentage, participant 2, 6 mos | 18.8
  REM percentage, participant 3, 6 mos | 9.7
  REM percentage, participant 4, 6 mos | 18.9
  REM percentage, participant 1, 12 mos | 18.2
  REM percentage, participant 2, 12 mos | 10.1
  REM percentage, participant 3, 12 mos | 27.5
  REM percentage, participant 4, 12 mos | 8.5
  REM percentage, participant 1, 18 mos | 27.8
  REM percentage, participant 2, 18 mos | 6
  REM percentage, participant 3, 18 mos | 19.8
  REM percentage, participant 4, 18 mos | 11.6

3. Other Pre Specified Outcome: An Exploratory Analysis Will Investigate Whether Normalization of REM Parameters Also Improves Other Measurements of Sleep Quality in Children With Autism.
Time Frame: 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Mullen Scales at 18 Months
Time Frame: 18 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Autism Diagnostic Observation Schedule (ADOS) at 6, 12 and 18 Months
Time Frame: 6, 12 and 18 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Vineland Parent Questionnaire at 3, 6, 12 and 18 Months
Time Frame: 3, 6, 12 and 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 18 months
Arm/Group | Open-Label Donepezil
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Study terminated due to lack of recruitment. No conclusions regarding the use of donepezil can be drawn from small sample size data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes